CLINICAL TRIAL: NCT00810355
Title: Effects of CBT and Cognitive Remediation on Work in Schizophrenia
Brief Title: Cognitive Behavior Therapy and Work Outcome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: Indiana University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: D6629-R
Record Dates: First submitted 2008-12-16; First posted 2008-12-18 (Estimated); Results first posted 2016-10-31 (Estimated); Last update posted 2017-05-23 (Actual); Status verified 2017-04

CONDITIONS: Schizophrenia
Keywords: Schizophrenia Spectrum Disorders; Cognitive Behavior Therapy; work
MeSH Terms: conditions — Schizophrenia | interventions — Self-Help Groups; Cognitive Behavioral Therapy; Cognitive Remediation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arm 1 (Active Comparator): Support group
  Interventions: Behavioral: Support Group
- Arm 2 (Experimental): Cognitive Behavior Therapy
  Interventions: Behavioral: Support Group; Behavioral: Cognitive Behavior Therapy
- Arm 3 (Experimental): Cognitive Behavior Therapy and Cognitive Remediation
  Interventions: Behavioral: Support Group; Behavioral: Cognitive Behavior Therapy; Behavioral: Cognitive Remediation

INTERVENTIONS:
Behavioral: Support Group — General support and problem solving for work activity
Behavioral: Cognitive Behavior Therapy — Individual and group therapy focused on identifying and correcting maladaptive beliefs about work
  Arms: Arm 2; Arm 3
Behavioral: Cognitive Remediation — Computerized training to enhance cognitive functioning.
  Arms: Arm 3

SUMMARY:
This research studies the effects of Cognitive Behavior Therapy and Cognitive Remediation on work for persons with schizophrenia. Cognitive Behavior Therapy is a form of counseling that helps people to improve their mental health by changing the way they think about themselves and others. Cognitive Remediation is an exercise to improve the thinking process. The purpose of this study is to determine the extent to which Cognitive Remediation combined with Cognitive Behavior Therapy helps people who are working.

DETAILED DESCRIPTION:
Objectives: The proposed grant seeks to compare the effects of a manualized form of Cognitive Behavior Therapy (CBT) combined with Cognitive Remediation (CR) with CBT alone and Support Services (SS) alone on vocational outcomes for persons with schizophrenia spectrum disorders. Key hypotheses are: I) Participants receiving CBT +CR will work more weeks and hours than participants receiving CBT alone or SS alone; II) Participants receiving CBT + CR condition will show better work performance than the CBT alone and SS alone conditions; III) Participants receiving CBT + CR will experience greater improvements in symptoms, dysfunctional beliefs and quality of life than the CBT alone or SS alone conditions Research Plan: One hundred twenty participants with Structured Clinical Interview for DSM-IV (SCID) confirmed diagnoses of schizophrenia or schizoaffective disorder will be recruited from the Roudebush VA Medical Center , surrounding mental health centers and the Marion VA Medical Center. Participants with these diagnoses will be eligible if they are sufficiently stable to sustain participant in rehabilitation, as defined by no hospitalizations, medication or housing changes in the last 30 days. Participants will be offered a 6 month paid job placement and randomly assigned to receive either CBT + CR, CBT only or SS only.

Methodology: Following informed consent, a baseline assessment will include an inventory of work, residential, substance abuse, legal, quality of life, psychiatric and service utilization history. Participants will be offered a 26-week job placement at the VA Medical center or within the community and randomly assigned to receive 6 months of either CBT +CR, CBT only or SS. Jobs will include entry-level positions supervised by regular job site supervisors. Participants in the SS condition will attend a weekly individual and support group offering unstructured support regarding work related problems they identify. Participants in the CBT group will attend weekly group and individual sessions employing a manualized CBT intervention to identify and correct dysfunctional cognitions related to work. Participants in the CBT + CR condition will attend meetings as indicated for CBT along with performing cognitive exercises on the computer, progressing at their own pace. Hours of work will be recorded weekly. Work performance will be measured biweekly. Symptoms and cognitions will be assessed every 2 months. Primary forms of data analyses will be multivariate repeated measure analyses of variance in which CBT +CR, CBT only and SS groups will be compared on vocational, symptom, and self-esteem variables.

Results: The investigators have recently demonstrated in separate randomized controlled trials that CBT and CR can be fully implemented in a VA setting and that each leads to better work outcomes in schizophrenia. Means and standard deviations of key outcomes have been determined and are used in the power analysis for this study.

Significance: The proposed research aims provide a scientifically sound exploration of the therapeutic value of productive activity in the rehabilitation of persons with schizophrenia and to determine the extent to which manualized CBT procedures when combined with CR may contribute to the success of this process. Results may provide exportable guidelines for augmenting work services with an appropriate psychological treatment. This information may lead to more effective rehabilitation programs as well as increases in productivity, functional independence and an enhanced quality of life for persons with schizophrenia. The study also fulfills the rehabilitation goal of maximum inclusion by providing CBT and CR services that may make it possible for some patients to function at work that otherwise could not.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of schizophrenia spectrum disorder,
* interest in vocational rehabilitation

Exclusion Criteria:

* No changes in medication type or housing in the last 30 days,
* mental retardation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2009-10-01 (Actual); Primary Completion 2015-08-06 (Actual); Study Completion 2015-08-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Lysaker, PhD, Principal Investigator — Richard L. Roudebush VA Medical Center, Indianapolis, IN
Locations (1):
- Richard L. Roudebush VA Medical Center, Indianapolis, IN, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 12 subjects consented, but failed to complete intake procedures for randomization. This is why the final results total enrollment number differs from the protocol enrollment number.
Groups:
- Cognitive Behavior Therapy and Cognitive Remediation: Support Group: General support and problem solving for work activity
  Cognitive Behavior Therapy: Individual and group therapy focused on identifying and correcting maladaptive beliefs about work
  Cognitive Remediation: Computerized training to enhance cognitive functioning.
Period: Overall Study
Arm/Group | Support Group | Cognitive Behavior Therapy | Cognitive Behavior Therapy and Cognitive Remediation
Started | 25 | 25 | 25
Completed | 11 | 8 | 14
Not Completed | 14 | 17 | 11
Not completed — Lost to Follow-up | 13 | 17 | 11
Not completed — Withdrawal by Subject | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Support Group: Support group
  Support Group: General support and problem solving for work activity
- Cognitive Behavior Therapy: Cognitive Behavior Therapy
  Support Group: General support and problem solving for work activity
  Cognitive Behavior Therapy: Individual and group therapy focused on identifying and correcting maladaptive beliefs about work
- Cognitive Behavior Therapy and Cognitive Remediation: Cognitive Behavior Therapy and Cognitive Remediation
  Support Group: General support and problem solving for work activity
  Cognitive Behavior Therapy: Individual and group therapy focused on identifying and correcting maladaptive beliefs about work
  Cognitive Remediation: Computerized training to enhance cognitive functioning.
- Total: Total of all reporting groups
Arm/Group | Support Group | Cognitive Behavior Therapy | Cognitive Behavior Therapy and Cognitive Remediation | Total
Number analyzed (Participants) | 25 | 25 | 25 | 75
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 23 | 25 | 25 | 73
  >=65 years | 2 | 0 | 0 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 1 | 4
  Male | 24 | 23 | 24 | 71
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 15 | 14 | 15 | 44
  White | 10 | 11 | 9 | 30
  More than one race | 0 | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 25 | 25 | 25 | 75

OUTCOME MEASURES:

1. Primary Outcome: Work Quality
Description: Average work performance scored on the Work Behavior Inventory (WBI) by total average of the 5 subscales. Scores range from 1-5. Higher scores represent better work performance.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Support Group | Cognitive Behavior Therapy | Cognitive Behavior Therapy and Cognitive Remediation
Number analyzed (Participants) | 25 | 25 | 25
scores on a scale | 3.01 (0.33) | 3.23 (.35) | 3.33 (.38)

2. Primary Outcome: Work Quantity
Description: Average number of hours worked per week. Higher numbers represent more hours worked, ranging from 0-40.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: hours worked per week
Arm/Group | Support Group | Cognitive Behavior Therapy | Cognitive Behavior Therapy and Cognitive Remediation
Number analyzed (Participants) | 25 | 25 | 25
hours worked per week | 14.79 (7.77) | 15.04 (6.56) | 17.73 (6.00)

3. Primary Outcome: Symptoms
Description: Symptoms (positive, negative, cognitive, hostility, and depression subscales) are rated on Positive and Negative Syndrome Scale (PANSS). These are averages of each subscale: positive (range 6-42), negative (range 8-56), cognitive (range 7-49), hostility (range 4-28), depression (range 4-28). Higher scores indicate more extreme /worse symptoms.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Support Group | Cognitive Behavior Therapy | Cognitive Behavior Therapy and Cognitive Remediation
Number analyzed (Participants) | 25 | 25 | 25
scores on a scale
  average positive symptoms | 17.79 (5.03) | 17.11 (4.48) | 15.85 (5.13)
  average negative symptoms | 20.97 (4.74) | 20.61 (4.84) | 19.42 (4.32)
  average cognitive symptoms | 18.44 (3.85) | 16.91 (3.37) | 16.46 (3.04)
  average hostility symptoms | 8.24 (2.79) | 7.09 (2.28) | 7.17 (2.54)
  average depression symptoms | 11.62 (2.95) | 11.86 (3.72) | 11.66 (3.60)

ADVERSE EVENTS:
Arm/Group | Support Group | Cognitive Behavior Therapy | Cognitive Behavior Therapy and Cognitive Remediation
Serious Adverse Events (participants affected / at risk) | 1/25 | 0/25 | 1/25
Other Adverse Events (participants affected / at risk) | 0/25 | 0/25 | 0/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Support Group (N=25) | Cognitive Behavior Therapy (N=25) | Cognitive Behavior Therapy and Cognitive Remediation (N=25)
psychiatric hospitalization (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1) — suicide ideation

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes